CLINICAL TRIAL: NCT04181567
Title: A Randomized, Double-blind, Comparison of the Efficacy, Safety, and Relapse of Electroconvulsive Therapy (ECT) to ECT Plus Agomelatine in the Treatment of Patients With Major Depressive Disorder
Brief Title: Comparison of the Efficacy, Safety, and Relapse of ECT to ECT Plus Agomelatine for Depressed Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ching-Hua Lin, MD, PhD, Chief of Adult Psychiatry, Kaohsiung Kai-Suan Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOST-103-2314-B-280-001-MY3; KSPH-2013-36 (Other: Kaohsiung Municipal Kai-Syuan Psychiatric Hospital)
Record Dates: First submitted 2019-11-24; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Major Depressive Disorder
Keywords: electroconvulsive therapy; agomelatine; relapse; major depressive disorder; response
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Electroconvulsive Therapy; agomelatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electroconvulsive therapy + agomelatine (Experimental): electroconvulsive therapy 2 times weekly + agomelatine 50 mg daily
  Interventions: Other: electroconvulsive therapy; Drug: agomelatine
- electroconvulsive therapy + placebo (Active Comparator): electroconvulsive therapy 2 times weekly + placebo
  Interventions: Other: electroconvulsive therapy; Drug: Placebo

INTERVENTIONS:
Other: electroconvulsive therapy — electroconvulsive therapy 2 times weekly
  Other Names: ECT
Drug: agomelatine — agomelatine
  Arms: electroconvulsive therapy + agomelatine
Drug: Placebo — placebo
  Arms: electroconvulsive therapy + placebo

SUMMARY:
Our hypothesis is that using antidepressants during the ECT has a better efficacy and longer time to relapse/recurrence to the ECT without antidepressants. The purpose of this study is to compare the efficacy, safety, and time to relapse/recurrence of ECT to ECT plus agomelatine in the treatment of patients with major depressive disorder. Inpatients with major depressive disorder for ECT will be randomly assigned to double-blind treatment with placebo or agomelatine 50 mg/d.

DETAILED DESCRIPTION:
Objective: Electroconvulsive therapy (ECT) is the safe and the most effective treatment for patients with major depressive disorder. It is still inconclusive whether antidepressants are continued during the course ot ECT. In terms of efficacy and safety, three essential questions arise: 1) does concomitant treatment improve the short-term antidepressant effects of ECT, 2) does concomitant treatment reduce the rate of early relapse/recurrence following ECT, 3) does concomitant treatment has more side effects? The purpose of this study is to conduct a clinical trial to compare the efficacy, safety, and time to relapse/recurrence of ECT to ECT plus agomelatine in the treatment of patients with major depressive disorder.

Methods: This is a prospective study. Inpatients with major depressive disorder for ECT will be randomly assigned to double-blind treatment with placebo or agomelatine 50 mg/d. After the ECT, the patients who meet the response criteria (i.e., at least a 50% reduction in symptom scores) or receive at least 6 treatments (i.e., acute phase) will receive the agomelatine 50 mg/d for 3 months (i.e., follow-up phase). The severity of depression, severity of anxiety, psychosocial functioning and side effects will be measured using the 17-item Hamilton Rating Scale for Depression (HAMD-17), the Clinical Global Impression-Severity (CGI-S), Depression and Somatic Symptoms Scale (DSSS), Zung's Depression Scale (ZDS), Hamilton Anxiety Rating Scale (HAM-A), Global Assessment of Functioning (GAF), Work and Social Adjustment Scale (WSAS), and UKU Side Effect Rating Scale before ECT, after every 3 sessions of ECT, at the end of acute ECT, and monthly during the 3-month follow-up period. Medical Outcomes Study Short-Form 36, Arizona Sexual Experiences Scale(ASEX), MINI Mental State Examination (MMSE), neuropsychological tests, and electroencephalography will be assessed before ECT, after ECT, and after the 3-month follow-up period. Questionnaire for patient attitudes about ECT after acute ECT will be completed. The Pearson chi-square test will be used to compare the response rate and remission (i.e., HAM-17≦7) rate between two groups. Analyses of group differences in efficacy will be performed by generalized estimating equations or ANCOVA. Survival analysis will be used to compare the time to response/remission and time to relapse/recurrence (i.e., HAM-D-17≧14 or CGI-S ≧4 or rehospitalization) after ECT between two groups.

Expected results: The results will provide evidence base for clinicians to decide to use antidepressants during ECT or not.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder
* Aged 18 years or older
* HAMD-17 >=18
* CGI-S >=4
* Treatment-resistant depression: a lack of response to two or more adequate trials of different classes of antidepressants
* Given written informed consent

Exclusion Criteria:

* History of schizophrenia, schizoaffective disorder or organic mental disorders
* Severe cognitive impairment
* Female subjects with lactation or pregnancy
* Serious medical conditions or neurological illnesses that restricte the use of ECT
* Receiving ECT within the 6 months
* Substance abuse/dependence within the 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Rating Scale for Depression (HAMD-17) | up to month 3.
  The HAMD-17 is widely used in clinical setting to evaluate depression symptoms in the past week. Higher total HAMD-17 scores (ranging from 0 to 52) indicate more severe depression.

SECONDARY OUTCOMES:
Clinical severity by Clinical Global Impression-Severity (CGI-S) | In acute phase, the CGI-S is rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination). In follow-up phase, the CGI-S is rated at months 1, 2, and 3.
  The CGI-S is developed for use in NIMH-sponsored clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI comprises one-item measures evaluating the severity of psychopathology from 1 to 7 and higher scores indicate higher severity.
Work and Social Adjustment Scale (WSAS) | In acute phase, the WSAS is rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination). In follow-up phase, the WSAS is rated at months 1, 2, and 3.
  The Work and Social Adjustment Scale (WSAS) is a 5-item self-rating scale designed to measure psychosocial functional impairment. Each item is scored from 0 (not affected at all) to 8 (severely affected).
UKU side effects rating scale | In acute phase, the UKU scale is rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination). In follow-up phase, the UKU scale is rated at months 1, 2, and 3.
  UKU side effects rating scale, with the score of each item ranging from 0 (none) to 3 (severe), is used to measure adverse events during the study period.
Electroencephalograph (EEG) | In acute phase, the EEG is recorded at baseline and again at week 6 (or on early termination). In follow-up phase, the EEG is recorded at month 3.
  The EEG is used to analyze the change of electroencephalogram complexity. EEG The recording lasted about 3 minutes after habituation to environment, and the EEG technician monitored subject vigilance. Recordings are in 19 electrodes (Fp1, Fp2, F7, F3, Fz, F4, F8, T7, C3, Cz, C4, T8, P7, P3, Pz, P4, P8, O1, O2) in the standard 10-20 International placement with mastoid reference. The raw EEG signal is transposed to MATLAB software (MathWorks Inc., Natick, MA, USA) for processing. Each electrode complexity will be calculated.
Medical Outcomes Study Short-Form 36 (SF-36) | In acute phase, the SF-36 is rated at baseline and again at week 6 (or on early termination). In follow-up phase, the SF-36 is rated at month 3.
  The SF-36 is used to assay the quality of life. Scores for the 8 SF-36 subscales range from 0 to 100, with a higher score representing better QOL.
Mini Mental State Examination (MMSE) | In acute phase, the MMSE is administered at baseline and again at week 6 (or on early termination). In follow-up phase, the MMSE is administered at month 3.
  The MMSE used to assay the cognitive function. It consists of 30 points. Lower scores indicate poorer performance and greater cognitive impairment. The total score ranges from 0 to 30.
Arizona Sexual Experiences Scale (ASEX) | In acute phase, the ASEX is rated at baseline and again at week 6 (or on early termination). In follow-up phase, the ASEX is rated at month 3.
  The ASEX is used to assay the sexual dysfunction. The ASEX taps five domains of sexual function using 6-point Likert scales scored from 1 (hyperfunction) to 6 (extreme hypofunction) to yield a total score ranging from 5 to 30.
Depression and Somatic Symptoms Scale (DSSS) | In acute phase, the DSSS is rated at baseline, and again at weeks 1, 2, 3, 4, 5 and 6 (or on early termination). In follow-up phase, the DSSS is rated at months 1, 2, and 3.
  The DSSS, a self-rating scale, is used to assay the severity of depression. The DSSS contains 22 items. Item responses are ranked from 0 to 3, with higher scores corresponding to more severe depression.
The Wechsler Memory Scale (WMS). | In acute phase, the WMS is administered at baseline and again at week 6 (or on early termination). In follow-up phase, The WMS is administered at month 3.
  The WMS is designed to measure different memory functions. Higher scores indicate higher memory functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Municipal Kai-Syuan Psychiatric Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin CH, Yang WC, Chan MH, Chen CC. The Relationship Between Depression and Pain During Acute Electroconvulsive Therapy and Follow-Up Period for Patients With Treatment-Resistant Depression. J ECT. 2022 Sep 1;38(3):192-199. doi: 10.1097/YCT.0000000000000830. Epub 2022 Mar 1. PMID 35220359